CLINICAL TRIAL: NCT00113139
Title: An Investigation to Examine a Telephone Based Stress Management and Coping Skills Intervention for Patients Waiting for Lung Transplant
Brief Title: Investigational Study of Psychological Intervention in Recipients of Lung Transplant (INSPIRE)
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00009150; R01HL065503 (NIH); 176
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-03

CONDITIONS: Lung Diseases; Depression
MeSH Terms: conditions — Lung Diseases; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone-based coping skills (Experimental): Telephone-based coping skills intervention
  Interventions: Behavioral: Telephone-based coping skills/stress management
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Telephone-based coping skills/stress management — Telephone-based coping skills/stress management: 12 weekly sessions.
  Other Names: Coping Skills Training (CST)
  Arms: Telephone-based coping skills
Other: Usual Care — Usual care participants continued their routine and usual treatments and do not receive the 12 telephone training sessions.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to examine the effectiveness of a telephone-based cognitive behavioral therapy intervention to alleviate psychological distress among lung transplant patients.

DETAILED DESCRIPTION:
BACKGROUND:

Lung transplantation is a relatively new procedure developed to increase life expectancy in selected individuals with irreversible end-stage lung disease. In the brief period since its inception, it appears that lung transplantation has achieved its initial aim of extending life. Despite these successes, lung transplantation remains fraught with difficult challenges for the patient and the medical community. The pre-surgical waiting period is a particularly stressful time. The long, uncertain wait for an organ, the marked decline in functional capacity, the tremendous financial burden, and the prospect of a complicated medical regimen after surgery, combine to exert a profound strain on patients' coping capacities. Not surprisingly, the rate of clinically significant psychological distress during this period is quite high, with rates of clinical depression, panic, anxiety and adjustment disorders far exceeding those observed in the general population. Although it is well established that brief, focused cognitive-behavioral therapy (CBT) can significantly improve psychological function in medically ill persons, the wide geographic distribution of transplant patients, along with their marked debilitation makes face-to-face delivery of such therapy extremely difficult. Recent pilot data have demonstrated the feasibility and short-term efficacy of a telephone-based psychological intervention with patients awaiting transplant.

DESIGN NARRATIVE:

INSPIRE was a collaborative study between Duke University Medical Center and Washington University Medical School. Participants first completed a baseline evaluation, including an interview with a staff member, tests of memory and concentration, and a questionnaire packet. They were then randomly assigned (by chance) to one of 2 groups: Stress Management (by phone) or Usual Care. Stress management participants received a phone call from an INSPIRE interventionist every week for 12 weeks; the phone sessions focused on helping to reduce stress and learning new skills to better cope with lung disease and the upcoming transplant. The INSPIRE staff interventionists were all psychologists who had been trained to work with patients with lung disease. Usual care participants continued their routine and usual treatments and did not receive the 12 telephone training sessions. Participants completed follow-up evaluations three months after the initial (baseline) evaluation, after transplant surgery, and twelve months after the initial evaluation. The primary outcome measures were measures of health-related quality of life, general psychological well-being, and social support.

ELIGIBILITY:
Inclusion Criteria:

* Potential lung-transplant candidates listed for lung transplantation at Duke University Medical Center or Washington University

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2000-09; Primary Completion 2007-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Survival/all-cause mortality | 6 months & 18 months post-transplant

SECONDARY OUTCOMES:
Quality of live | 6 months & 18 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: James A Blumenthal, Ph.D, Principal Investigator — Duke University Medical Center, Dept of Psychiatry & Behavioral Sciences

REFERENCES:
- [Background] Napolitano MA, Babyak MA, Palmer S, Tapson V, Davis RD, Blumenthal JA; Investigational Study of Psychological Intervention in Recipients of Lung Transplant (INSPIRE) Investigators. Effects of a telephone-based psychosocial intervention for patients awaiting lung transplantation. Chest. 2002 Oct;122(4):1176-84. doi: 10.1378/chest.122.4.1176. PMID 12377839
- [Background] Parekh PI, Blumenthal JA, Babyak MA, LaCaille R, Rowe S, Dancel L, Carney RM, Davis RD, Palmer S; INSPIRE Investigators. Gas exchange and exercise capacity affect neurocognitive performance in patients with lung disease. Psychosom Med. 2005 May-Jun;67(3):425-32. doi: 10.1097/01.psy.0000160479.99765.18. PMID 15911906
- [Background] Parekh PI, Blumenthal JA, Babyak MA, Merrill K, Carney RM, Davis RD, Palmer SM; INSPIRE Investigators. Psychiatric disorder and quality of life in patients awaiting lung transplantation. Chest. 2003 Nov;124(5):1682-8. doi: 10.1378/chest.124.5.1682. PMID 14605035
- [Derived] Smith PJ, Blumenthal JA, Carney RM, Freedland KE, O'Hayer CVF, Trulock EP, Martinu T, Schwartz TA, Hoffman BM, Koch GG, Davis RD, Palmer SM. Neurobehavioral functioning and survival following lung transplantation. Chest. 2014 Mar 1;145(3):604-611. doi: 10.1378/chest.12-2127. PMID 24233282